CLINICAL TRIAL: NCT05525143
Title: Incidence and Risk Factors of Postpartum Hemorrhage at the Brugmann University Hospital in Comparison to the Literature
Brief Title: Postpartum Hemorrhage: Incidence and Risk Factors
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of department, anesthesiology, Brugmann University Hospital
Other Study IDs: PPH
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pregnant women who have given birth vaginally or by cesarean section — Full-term pregnant women who have given birth vaginally or by cesarean section with PPH. Descriptive statistics and possible causal factors

SUMMARY:
Postpartum hemorrhage(PPH) is a major cause of maternal morbidity and mortality across the world. Incidence of PPH varies in the literature from 2 to 10%, most recent studies find around 10% of PPH and 2% of severe PPH.

In this study, the incidence of PPH in the maternal ward of the CHU Brugmann will be analyzed. This is a tertiary maternal ward with a high proportion of high risk pregnancies with around 3000 admissions per year.

Primary aim of this study is to evaluate the epidemiology of PPH in the CHU Brugmann, incidence and possible underlying causes will be identified and compared to the current literature. A data mining technique will be used to construct a prediction model for PPH.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have given birth vaginally or by cesarean section at the CHU Brugmann between January 1, 2020 and August 31, 2022
* ≥ 18 years

Exclusion Criteria:

* Age ≤ 18 years
* Age > 60 years
* delivery before 25th week of pregnancy
* delivery outside of the hospital
* abortion

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women who have given birth vaginally or by cesarean section
Study Population: Pregnant women who have given birth vaginally or by cesarean section at the CHU Brugmann between January 1, 2020 and August 31, 202
Sampling Method: Non-Probability Sample
Enrollment: 2402 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of PPH | 48 hours
  Descriptive statistics of incidence (%) of PPH occuring during the first 48h after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Besse, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deneux-Tharaux C, Bonnet MP, Tort J. [Epidemiology of post-partum haemorrhage]. J Gynecol Obstet Biol Reprod (Paris). 2014 Dec;43(10):936-50. doi: 10.1016/j.jgyn.2014.09.023. Epub 2014 Nov 6. French. PMID 25447386
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Reale SC, Easter SR, Xu X, Bateman BT, Farber MK. Trends in Postpartum Hemorrhage in the United States From 2010 to 2014. Anesth Analg. 2020 May;130(5):e119-e122. doi: 10.1213/ANE.0000000000004424. PMID 31567319
- [Background] Diaz V, Abalos E, Carroli G. Methods for blood loss estimation after vaginal birth. Cochrane Database Syst Rev. 2018 Sep 13;9(9):CD010980. doi: 10.1002/14651858.CD010980.pub2. PMID 30211952
- [Background] Nyflot LT, Sandven I, Stray-Pedersen B, Pettersen S, Al-Zirqi I, Rosenberg M, Jacobsen AF, Vangen S. Risk factors for severe postpartum hemorrhage: a case-control study. BMC Pregnancy Childbirth. 2017 Jan 10;17(1):17. doi: 10.1186/s12884-016-1217-0. PMID 28068990
- [Background] Girault A, Deneux-Tharaux C, Sentilhes L, Maillard F, Goffinet F. Undiagnosed abnormal postpartum blood loss: Incidence and risk factors. PLoS One. 2018 Jan 10;13(1):e0190845. doi: 10.1371/journal.pone.0190845. eCollection 2018. PMID 29320553
- [Background] Anger H, Durocher J, Dabash R, Winikoff B. How well do postpartum blood loss and common definitions of postpartum hemorrhage correlate with postpartum anemia and fall in hemoglobin? PLoS One. 2019 Aug 22;14(8):e0221216. doi: 10.1371/journal.pone.0221216. eCollection 2019. PMID 31437195
- [Background] Goad L, Rockhill K, Schwarz J, Heyborne K, Fabbri S. Development and validation of a prediction model for postpartum hemorrhage at a single safety net tertiary care center. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100404. doi: 10.1016/j.ajogmf.2021.100404. Epub 2021 May 25. PMID 34048966
- [Background] Ambler G, Omar RZ, Royston P. A comparison of imputation techniques for handling missing predictor values in a risk model with a binary outcome. Stat Methods Med Res. 2007 Jun;16(3):277-98. doi: 10.1177/0962280206074466. PMID 17621472